CLINICAL TRIAL: NCT05135390
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of HSK21542 Injection in Maintenance Hemodialysis Patients with Chronic Kidney Disease-associated Pruritus
Brief Title: A Clinical Trial Evaluating the Efficacy and Safety of HSK21542 in Patients with Chronic Kidney Disease-Associated Pruritus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK21542-302
Record Dates: First submitted 2021-11-15; First posted 2021-11-26 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Pruritus; Hemodialysis Patients with Moderate-to-Severe Pruritus
Keywords: Hemodialysis Patients with Moderate-to-Severe Pruritus; HSK21542
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HSK21542 (Experimental): 0.3 μg/kg
  Interventions: Drug: HSK21542
- Placebo (Experimental): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK21542 — three times per week
  Arms: HSK21542
Drug: Placebo — three times per week
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled study. About 544 maintenance hemodialysis patients with moderate or above chronic kidney disease-associated pruritus are planned to be enrolled. They will randomized into the treatment group (HSK21542, 0.3 μg/kg) and the control group (placebo) at a 1:1 ratio.

DETAILED DESCRIPTION:
Double-blind Phase The Double-blind Phase of the study will consist of a 28-day Screening Visit, a 7-day Run-in Period, a 12 week Double-blind Treatment Period, and one week Follow-up Period. Informed consent will be obtained prior to performing any study-specific procedures. The Screening Visit will occur within 7 to 28 days prior to randomization to assess eligibility.

Open-label Extension Phase Patients who medication compliance ≥ 80% during the 12-week Double-blind Treatment Period and continue to meet other eligibility criteria will have the option to receive open label HSK21542 for an additional 40 weeks. The Open-label Extension Phase will be comprised of the Open-label Treatment Period and the Follow-up Period.

The last dose of open-label study drug will be administered at the last dialysis visit on Week 40, or Early Termination. A final safety Follow up Visit will be conducted 5-9 days after the End of Treatment/Early Termination Visit.

ELIGIBILITY:
The double-blind phase Inclusion Criteria:

1. Subjects who are willing to sign an informed consent form, fully understand the objectives and significance of the trial, and are willing to comply with the trial protocol before any of the study-related procedures start;
2. Aged ≥ 18 years old, male or female;
3. Patients with end-stage renal disease, who have received regular hemodialysis (including hemodiafiltration) 3 times per week for at least 3 months prior to screening (the judgment of regular hemodialysis is subject to the joint medical comment of the investigator and the sponsor);
4. Dry weight at screening: 40.0-135.0 kg (inclusive);
5. On different days of hemodialysis within 6 months prior to administration, at least two occurrences of single-pool urea clearance index (sp Kt/V) ≥ 1.2 or at least two occurrences of urea reduction ratios (URR) ≥ 65%, or one occurrence of sp Kt/V ≥ 1.2 and one occurrence of URR ≥ 65%;
6. Having completed at least 5 assessments of the Worst Itch Numeric Rating Scale from the lead-in period through D-1 and meeting the criteria of baseline itch intensity > 5 (defined as the average of all non-missing scores from the lead-in period to D-1; scores 0-10 indicates the range from no itch to the worst imaginable itch);
7. Male subjects who agree to use condoms in sexual intercourse during the study and within 3 months after the last dose; female subjects who have been menopausal for at least one year, or who have been sterilized permanently (e.g., fallopian tube occlusion, hysterectomy, bilateral salpingectomy); or women of childbearing potential who agree to take effective contraceptive measures during the study and within 3 months after the last dose, such as oral contraceptives, condoms, and contraceptive films.

The 0pen-label extension phase Inclusion Criteria：

1. Dry weight ≥ 40 kg;
2. Complete a double-blind study with medication adherence of ≥ 80%.

The double-blind phase Exclusion Criteria:

Exclusion criteria (those who meet any of the followings are ineligible):

1. Expecting to undergo renal transplantation and/or parathyroidectomy during the study，or parathyroid hormone >800 pg/mL;
2. Having a history of allergy to opioids, such as urticaria (Note: adverse effects related to opioid use, such as constipation and nausea, are not included as the exclusion criteria in this study);
3. Having used opioids within 7 days before screening, or being unable to avoid the use of opioids other than the investigational drug during the study;
4. Having participated in any clinical trial of other drug or medical device within 1 month before screening (received study medication or treated by the medical device in the clinical trial);
5. New or change of treatment received for hemoperfusion regimen within 3 months prior to screening or anticipating to adjust hemoperfusion regimen during the study;
6. Upper extremity blood pressure in a supine position during screening: systolic blood pressure < 90 mmHg, or diastolic blood pressure < 60 mmHg, or systolic blood pressure > 180 mmHg, or diastolic blood pressure > 110 mmHg;
7. Alanine transaminase (ALT) or AST (aspartate transaminase) > 2.5 × upper limit of normal (ULN), or total bilirubin > 2 × ULN at screening;
8. Blood sodium > 155 mmol/L at screening;
9. Hemoglobin < 80 g/L at screening;
10. Positive for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), syphilis antibody, or human immunodeficiency virus (HIV) antibody at screening;
11. Pruritus that may or must not be caused by ESRD or its complications (e.g., patients with pruritic dermatosis or cholestatic liver disease will be excluded);
12. New or change of treatment received including antihistamines (oral, intravenous, or topical), systemic or topical corticosteroids (except for otic or ophthalmic preparations) , calcium regulated phosphatase inhibitors, gabapentin, pregabalin, and other combination drugs that are restricted in 5.5.1, or whose treatment regimen must be changed during the expected double-blind study periodwithin 7 days prior to screening or anticipating inevitable treatment regimen adjustment during the study;

14. New or change of medications that may affect the judgment of antipruritic efficacy, including but not limited to antipsychotics, sedative-hypnotics, selective serotonin reuptake inhibitors (SSRIs), anxiolytics, or tricyclic antidepressants within 14 days prior to screening or anticipating inevitable treatment regimen adjustment during the study; 15. Females who are pregnant or breastfeeding; 16. Any physiological or psychological diseases or conditions that may increase the risk of the trial, affect the subject's compliance with the protocol, or affect the subject's completion of the trial, as judged by the investigator, including but not limited to:

1. Local pruritus limited to palms only;
2. Pruritus during hemodialysis only;
3. History of known or suspected abuse of or dependence on alcohol, narcotics or other drugs within 12 months before screening;
4. Severe systolic or diastolic heart failure within 6 months prior to screening, e.g., NYHA Class IV congestive heart failure (see Appendix 7 for NYHA functional classification criteria);
5. Severe mental illness or cognitive impairment (e.g., dementia);
6. Any other relevant acute or chronic neurological or psychiatric condition within 3 months prior to screening that, at the discretion of the investigator, is not suitable for enrollment (e.g., encephalopathy, coma, delirium);
7. Patients with malignancy, but excluding: curable cervical carcinoma in situ, skin basal cell or squamous cell carcinoma, or any other tumors that have been cured (no evidence of disease recurrence within 5 years).

The 0pen-label extension phase Exclusion Criteria:

1. During the double-blind treatment period, an adverse event occurred that may affect the subject's continued receipt of the study drug;
2. As determined by the investigator, there are any physical or psychological diseases or conditions that may increase the risk of the trial, affect the subject's compliance with the protocol, or affect the subject's completion of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 545 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with an improvement of ≥ 4 points from baseline in the weekly average of the daily Worst Itch Numeric Rating Scale (WI-NRS) after 12 weeks of treatment. | week 12
  In the NRS score, 0-10 represents different degrees of itching, the larger the number, the more severe the itching

SECONDARY OUTCOMES:
Change from baseline in subjects' quality of life (evaluated using the Skindex-10 scale ) after 12 weeks of treatment. | week 12
  The Skindex-10 Scale is a multidimensional questionnaire which assesses itch-related quality of life over the past week. The questions cover 3 domains: symptoms, emotions, and functioning domain. A lower total score represents better quality of life.
Change from baseline in subjects' quality of life (evaluated using the 5-D itch scale) . | Double-blind Phase：week 12,；Open-label Extension Phase: week 24, 40
  The 5-D Itch Scale is a multidimensional questionnaire which assesses itch-related quality of life over the past 2 weeks. The questions cover five dimensions of itch including the degree, duration of itch/day, direction (improvement/worsening), disability (impact on activities such as work), and body distribution of itch. A lower total score represents better quality of life.
Proportion of subjects with an improvement of ≥ 3 points from baseline in the weekly average of the daily Worst Itch Numeric Rating Scale (WI-NRS) after 12 weeks of treatment. | week 12
  In the NRS score, 0-10 represents different degrees of itching, the larger the number, the more severe the itching

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhong Da Hospital Southeast University, Nanjing, Jiangsu
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu BC, Li ZL, Zhang P, Zhong AM, Bai YL, Xu Y, Gao BH, Li YL, Wang Y, Zhou LH, Yao L, Wang JX, Yan R, Wang L, Liao B, Xie DQ, Yi XM, Guan TJ, Wang CL, Li GS, Li FQ, Chen JH; Anrikefon-302 study collaborator group. Efficacy and safety of anrikefon in patients with pruritus undergoing haemodialysis: multicentre, double blind, randomised placebo controlled phase 3 trial. BMJ. 2025 Aug 19;390:e085208. doi: 10.1136/bmj-2025-085208. PMID 40829896